CLINICAL TRIAL: NCT03615196
Title: Evaluation of USB005 in a Phase 1 Normal, Healthy Volunteer Ocular Safety and PK Study
Brief Title: Study of the Safety of USB005 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Biotest, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USB005-2017-01
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteers
Keywords: NorLeu3-A(1-7); USB005; aclerastide; corneal repair; corneal injury
MeSH Terms: conditions — Corneal Injuries | interventions — aclerastide; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- USB005 0.03% (Experimental): USB005 (aclerastide) Ophthalmic Solution 0.03%; single eye drop instillation three times a day to one eye during a 28-day treatment period (84 treatments)
  Interventions: Drug: USB005 (aclerastide) Ophthalmic Solution
- USB005 0.1% (Experimental): USB005 (aclerastide) Ophthalmic Solution 0.1%; single eye drop instillation three times a day to one eye during a 28-day treatment period (84 treatments)
  Interventions: Drug: USB005 (aclerastide) Ophthalmic Solution
- USB005 0.3% (Experimental): USB005 (aclerastide) Ophthalmic Solution 0.3%; single eye drop instillation three times a day to one eye during a 28-day treatment period (84 treatments)
  Interventions: Drug: USB005 (aclerastide) Ophthalmic Solution
- USB005 0.45% (Experimental): USB005 (aclerastide) Ophthalmic Solution 0.45%; single eye drop instillation three times a day to one eye during a 28-day treatment period (84 treatments)
  Interventions: Drug: USB005 (aclerastide) Ophthalmic Solution
- USB005 Placebo (Placebo Comparator): USB005 Ophthalmic Solution Placebo; single eye drop instillation three times a day to one eye during a 28-day treatment period (84 treatments)
  Interventions: Drug: USB005 Ophthalmic Solution Placebo

INTERVENTIONS:
Drug: USB005 (aclerastide) Ophthalmic Solution — Aclerastide ([Nle3]-Angiotensin II (1-7)) is aseptically formulated in USB005 Ophthalmic Solution for topical ophthalmic administration. Active pharmaceutical ingredient (API) levels ranging from 0.03% to 0.45% are formulated in a sterile vehicle consisting of 0.06% Sodium Phosphate Monobasic Anhydrous, USP; 3% Glycerol, USP; 1.4% Polyvinyl Alcohol, USP; and 0.5% Hydroxyethylcellulose (HEC 250 HHX), NF in Sterile Water for Injection, USP.
  Arms: USB005 0.03%; USB005 0.1%; USB005 0.3%; USB005 0.45%
Drug: USB005 Ophthalmic Solution Placebo — A clinical placebo formulated with the same excipients and packaged in the same container closure system as the active product, USB005 (aclerastide) Ophthalmic Solution.
  Arms: USB005 Placebo

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics of USB005 (aclerastide) Ophthalmic Solution.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, randomized, double-masked, placebo-controlled, multiple ascending dose study in healthy volunteers. Thirty-two male and female volunteer subjects, between the ages of 18 and 64 years of age, will be enrolled. Subjects will be enrolled in four dose-escalating cohorts of eight subjects and randomized to USB005 or placebo in a ratio of 3:1. Cohorts will be enrolled sequentially starting at the lowest concentration. The four cohorts will be identified as: Cohort 1(0.03% USB005 or placebo), Cohort 2 (0.1% USB005 or placebo), Cohort 3 (0.3% USB005 or placebo), and Cohort 4 (0.45% USB005 or placebo). Volunteers in the four cohorts will self-administer a single drop of USB005 or placebo into the study eye, three times a day for 28 days. The study eye in which the drug is applied to will be determined based on screening assessments. Subjects will be followed for 8 days after the last USB005 or placebo administration.

The safety and tolerability of USB005 will be demonstrated by local toxicity, adverse events, laboratory assessments, vital signs, and a comprehensive eye exam. Plasma samples will be taken at various time points throughout the study to characterize the pharmacokinetics of USB005. Dropouts will be replaced after consultation with the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers, aged 18-64 years (inclusive) at the time of signing the ICF;
2. For females:

   1. Surgically sterilized (eg, hysterectomy or bilateral oophorectomy) for at least 6 months prior to screening or postmenopausal (postmenopausal women must have no menstrual bleeding for at least 1 year prior to screening and menopause will be confirmed by a plasma FSH level of >40 IU/L) or
   2. Women of childbearing potential must be non-lactating and agree to use a highly effective acceptable form of birth control (e.g., established hormonal birth control plus a barrier method, double barrier method: intrauterine device plus condom or spermicidal gel plus condom) from 21 days prior to dosing until 7 days after dosing, and
   3. Women with a negative pregnancy test (β-hCG assay) at screening and Day -1;
3. Weight of 45-100 kg and BMI of 17.5-35 kg/m2 (inclusive);
4. Blood pressure no greater than 120/80 mm Hg (inclusive);
5. Healthy, as determined by medical history, physical examination, vital signs, and clinical laboratory tests, unless the Investigator considers an abnormality to be clinically irrelevant;
6. IOP measurement oculus uterque (OU, both eyes) <21 mm Hg at screening and Day -1;
7. BCVA 20/30 or better (LogMAR and Snellen Equivalent) at both the screening visit and Day -1 in at least 1 eye;
8. Normal vision as determined by comprehensive ocular examination;
9. Able and willing to provide signed, written, informed consent;
10. Willing to communicate with the Investigator and site staff and comply with all study procedures and requirements;
11. Willing and able to be confined to the clinical study site as required by the protocol.

Exclusion Criteria:

1. Any history of severe ocular trauma in either eye at any time;
2. Any history of previous intraocular or ocular laser surgery within the past 3 months or any refractive surgery procedure within the past 6 months of the screening visit in either eye;
3. Any condition preventing reliable ocular assessment (eg, applanation tonometry, fundus examination) in either eye;
4. Intended use of contact lenses during this study or 1 week before Day -1;
5. Current or chronic history of ocular disease within the past 3 months of screening visit in either eye;
6. Current or chronic history of ocular infection (bacterial, viral or fungal) or corneal irritation within the past 3 months of screening visit in either eye OR ongoing or recurrent ocular inflammation (ie, moderate to severe blepharitis, allergic conjunctivitis, peripheral ulcerative keratitis, scleritis, uveitis) in either eye;
7. Abnormal tearing, OR expected regular use of prescription or expected use of OTC tear substitutes within 4 weeks prior to Day -1, and for the duration of the study;
8. Previous or expected use of ocular (topical, periocular, intravitreal), local (inhaled or nasal), or systemic steroid or glucocorticoid medications within 4 weeks prior to Day -1, and for the duration of the study;
9. At the ophthalmic investigator's discretion, any volunteers who have a history of any significant ocular conditions in either eye that would contraindicate the use of the study medication, or that might affect the study conduct, or the interpretation of the study results;
10. Use of any non-diagnostic topical ophthalmic solutions through the duration of the study;
11. Clinically significant metabolic disease such as diabetes, asthma, or hypertension (ie, blood pressure >120/80 mm Hg on two successive visits during screening);
12. Taken any nicotine-containing products in the last 6 months prior to dosing or for the duration of the study;
13. At the Investigator's discretion, any volunteers with a history or presence of clinically significant cardiovascular disorders, including a history of orthostatic hypotension, arrhythmia and syncope (including vasovagal syncope), or respiratory, metabolic, renal, hepatic, immunologic, endocrine, dermatologic, venereal, hematologic, neurologic, psychiatric (eg, major depression with suicidal ideation, or suicide attempt), malignant neoplasm, musculoskeletal, connective tissue, urinary disease or disorders;
14. History of clinically significant drug or food allergy;
15. Positive HIV, hepatitis B or C viral test at screening;
16. Taken any prescription drugs within 14 days or within 5 half-lives, whichever is longer, prior to dosing;
17. Taken any non-prescription or OTC drugs including vitamins or herbal medications within 14 days or within 5 half-lives whichever is longer, prior to dosing;
18. History or presence, as judged by the Investigator, of drug or alcohol abuse (ie, alcohol consumption >2 drinks/day over the last 3 months prior to screening); drug abuse is any use of illegal drugs or prescription-drug over usage or addiction. A positive drug screen or alcohol screen will disqualify a volunteer from study participation;
19. Donated >400 mL and/or received any blood or blood products within the previous 3 months prior to screening;
20. Taken any investigational medication and/or participated in any clinical studies within 30 days of screening;
21. Any volunteer who, in the judgment of the Investigator, may not be able to cooperate fully with the study staff, may have difficulty following some study requirements, or is otherwise not qualified for the study;
22. Any volunteer who is directly involved in the conduct of the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Percentage of volunteers with dose limiting toxicities in each cohort | 36 days
Percentage of volunteers in each cohort with ocular adverse events | 36 days
Percentage of volunteers in each cohort with systemic adverse events | 36 days
Percentage of volunteers with clinically significant out of range laboratory values | 36 days

SECONDARY OUTCOMES:
Maximum observed concentrations (Cmax) | 36 days
Time to reach maximum observed plasma concentration (Tmax) after multiple ascending dose | 36 days
Apparent terminal half-life (T1/2) after multiple ascending dose | 36 days
Area under the plasma concentration versus time curve from time 0 to infinity (AUCinf) | 36 days
Area under the plasma concentration versus time curve up to the last measurable concentration (AUC0-last) | 36 days
Apparent clearance (CL/F) | 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sheety, MD, Principal Investigator — WCCT Global, Inc.
Locations (1):
- WCCT Global, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdallah WF, Louie SG, Zhang Y, Rodgers KE, Sivok E, S diZerega G, Humayun MS. NorLeu3A(1-7) Accelerates Clear Corneal Full Thickness Wound Healing. Invest Ophthalmol Vis Sci. 2016 Apr 1;57(4):2187-94. doi: 10.1167/iovs.15-18515. PMID 27116546